CLINICAL TRIAL: NCT01002638
Title: The Occlusive Dressing: a Comparative Randomized Trial on 2 Procedures of Treatment of Fingertips Traumatic Amputations
Brief Title: The Occlusive Dressing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulty
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4436
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Fingertips Traumatic Amputations
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Occlusive Dressing (Experimental)
  Interventions: Other: TEGADERM®
- Surgery (Active Comparator)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Other: TEGADERM® — It consists of the occlusive application of two Tegaderm®, a plastic dressing
  Arms: Occlusive Dressing
Procedure: Surgery — It consists of pulp reconstruction by a flap (for example palmar V-Y advancement flaps of Atazoy).
  Arms: Surgery

SUMMARY:
Fingers amputations are very common injuries among the patients arriving at the Emergency Department. Fingertips amputations classified in 2nd and 3rd zones, in accordance with Rosenthal's classification (after the solum unguis), constitute a large proportion of them. The treatment aims at restoring a pulp with its sensitivity and a good subcutaneous fat tissue. The usual care of these amputations is a surgical treatment: it consists of pulp reconstruction by a flap (for example palmar V-Y advancement flaps of Atazoy). These technique involve hospital admission, brachial plexus anaesthesia, a surgical approach with cicatrix and donor site morbidities, postoperative cares, post-surgical pain management. And of course attention must be paid to the risks of postoperative complications related either to anaesthesia and/or to surgery, like necrosis, infection, and others. We have developed a nonoperative treatment for fingertips amputations: the occlusive dressing. It's a technique that has been known for about twenty years, and that is currently developed by the teams SOS main of Professor Liverneaux in Strasbourg and of Professor Obert in Besançon. It consists of the occlusive application of two Tegaderm®, a plastic dressing. Then the finger macerates in an anaerobic medium, and could develop an uncomfortable smell induced by maceration process. The first results described by the preclinical studies of these two groups look satisfying on both the functional aspect (sensibility) and the aesthetic component (preservation of the finger length and curve), as well as for healing that occurs without infection. Moreover, the length of the treatment is of about only three or four weeks, and its cost is very low by comparison with the cost of the surgery itself. Nevertheless this technique is still not very common, and it has been reported in only five references in the literature [Mennen & Al., Farrell & Al., Lee & Al., Allen & Al., Tago Hiroyuk & Al.]. On the other hand, the mechanism of action and/or the active components of this occlusive dressing have not yet been the objects of extended studies. An explanatory hypothesis is that some anaerobic germs and/or growth factors might play an active role in the process. However, they have not been identified yet. The aim of our study is to validate through clinical and biological criteria this non operative method and to compare with surgical treatment. The study will be held in the Hand Department of the University Hospital of Strasbourg, under the direction of the Pr Liverneaux. It will imply the collaboration of the laboratory of medical bacteriology directed by Pr Piemont, and the research department of INSERM (Parogène laboratory) will focus on the biochemistry. From a clinical point of view, a certain number of objective functional criteria will be measured: the pain will be evaluated by a visual analogic scale and the DN4 scale; the functional disability will be measured with the french version of the Disability Arm Shoulder Hand of Dubert; the pulpar 3D volume will be calculated from the numerical pictures with a computerized file, the cutaneous depth will be measured by 3D U.S; the tactile sensibility will be tested by standardized monofilaments and Weber's test and the dermatoglyphics of both handsides will be compared. In addition, the subjective feeling of the patients will be recorded through a visual and analogical scale of satisfaction. The purpose of the biological component of the study will be to put into light and to identify the components that are active in the process. This will be performed by the direct examination and by bacteriological cultures, and will look for the anaerobic, aerobic germs and the yeasts.The biochemical studies will first include a non specific search of growth factors, cytokines and interleukins. In a second step, specific researches will be undertaken if necessary in accordance with the results of the first investigations. By this study, the investigators would like to scientifically confirm the efficiency of this method with objective as well as subjective criteria, and to identify the underlying biomechanisms of the process.

DETAILED DESCRIPTION:
This is a multicentre, randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Fingertips traumatic amputations (zone 2 or 3)

Exclusion Criteria:

* Fingertips traumatic amputations (zone 1 or 4)
* Fingertips amputations non traumatic
* Traumatic history on the finger,, nervous traumatism or nerve tumor on the same upper limb
* Nervous tumor history or cervical spine traumatism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
the tactile sensibility will be tested by standardized monofilaments | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: philippe LIVERNEAUX, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (3):
- France (3):
  - University Hospital, Besançon
  - University Hospital, Bordeaux
  - University Hospital, Strasbourg